CLINICAL TRIAL: NCT03958240
Title: Deciphering Mechanisms Underlying Cancer Immunogenicity
Acronym: DECIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19 GENE 13
Record Dates: First submitted 2019-05-20; First posted 2019-05-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer; Ovarian Cancer; Cervical Cancer; Cervical Intraepithelial Neoplasia 3; Glioblastoma Multiforme of Brain Stem; Non Small Cell Lung Cancer; Anal Cancer
Keywords: Head and Neck Cancer; Ovarian Cancer; Cervical Cancer; Cervical Intraepithelial Neoplasia 3; Glioblastoma Multiforme of Brain Stem; Non Small Cell Lung Cancer; Anal Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Non-Small-Cell Lung; Anus Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with local and/or metastatic solid malignant tumor (Other): Patient receiving an anticancer treatment in the context of their standard care.
  Interventions: Other: Blood samples, tumor biopsy specimens and ascites samples will be collected.

INTERVENTIONS:
Other: Blood samples, tumor biopsy specimens and ascites samples will be collected. — Blood samples, tumor biopsy specimens and ascites samples will be collected at different time points (if feasible, according to the samples taken in the standard practice) for a maximum follow-up period of 5 years from baseline:
  * at Baseline.
  * at every surgical procedure or tumor biopsy.
  * every 6 months (± 2 months) (only blood sample).
  * at the time of the progression or recurrence, additional samples will be collected, and optionally at the time of the following progressions or recurrences (if applicable).
  For patients undergoing a RT treatment, blood samples will be collected before the RT (i.e. at the time of planning CT-scan), at the last session of RT (± 2 days) and 3 months after the end of the RT (± 2 weeks).

SUMMARY:
This trial is a translational, open-label, multicentric, prospective cohort study of 1100 patients aiming to describe the PD-1 (programmed death) expression in T cells (T lymphocytes) in different solid tumors.

The study will be conducted on a population of patients with local and/or metastatic malignant solid tumor and who are followed within a standard of care procedure or clinical trial.

Patients with any of the following tumor types may be enrolled in the trial:

* Head and neck cancer,
* Ovarian cancer,
* Cervical cancer,
* Pre-invasive CIN III cervical cancer (Cervical Intra-epithelial Neoplasia III cervical cancer),
* Other solid tumor types (including glioblastoma, NSCLC (Non-small cell lung cancer), anal cancer)

Each tumor type will be considered as an independent cohort.

For each included patient, biological specimen (tumor sample, blood samples and ascites samples if applicable) will be collected.

Study participation of each patient will be 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histologically documented local or metastatic solid malignant tumor (head and neck, ovarian, cervical, and other tumor types including, but not limited to glioblastoma, NSCLC and anal cancer) or patients with pre-invasive cervical high grade dysplasia (CIN II or III)
2. Age ≥ 18 years at the time of study entry
3. Patient followed within a standard of care procedure or clinical trial
4. ECOG Performance status 0-2
5. Patient able to participate and willing to give informed consent prior performance of any study-related procedures and to comply with the study protocol
6. Patient affiliated to a Social Health Insurance in France
7. Patient may participate to other clinical trials

Exclusion Criteria:

1. Known history of positive test for Hepatitis B virus or Hepatitis C virus or Immunodeficiency Virus (HIV) or Hanta virus
2. Any condition contraindicated with blood sampling procedures required by the protocol (including Hemoglobin < 8g/dl)
3. Patient pregnant, or breast-feeding
4. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure
5. Patient who has forfeited his/her freedom by administrative or legal award or who is under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2020-01-17 (Actual); Primary Completion 2033-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of CD4 and CD8 T cells expressing PD-1 | 5 years for each patient

SECONDARY OUTCOMES:
Rate of patients presenting a high Trm (Tissue resident memory) infiltrate in tumor samples | 5 years for each patient

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hopital Larrey, Toulouse
  - Hopital Rangueil, Toulouse
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse